CLINICAL TRIAL: NCT04997915
Title: Acute Kidney Injury in COVID-19 Patients Admitted to the ICU: a Multicenter Cohort Analysis in 9 Large Hospitals in Belgium
Brief Title: Acute Kidney Injury in Coronavirus Disease-19 (COVID-19) Patients Admitted to the Intensive Care Unit (ICU)
Acronym: COVID-AKI-B
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); University Hospital, Antwerp (Other); Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other); General Hospital Groeninge (Other); AZ Delta (Other); AZ Turnhout (Other); AZ Sint-Jan AV (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08285
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-01

CONDITIONS: Critical Illness; COVID-19 Pneumonia; Acute Kidney Injury
Keywords: Acute kidney injury; COVID-19; ICU; Epidemiology; Kidney Replacement Therapy; Acute Kidney Disease; Recovery; Mortality; Survival
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical COVID-19: Critical COVID-19 patients admitted to the ICU
  Interventions: Other: Observational study exploring the epidemiology and outcomes of AKI in critical COVID-19 patients admitted to the ICU

INTERVENTIONS:
Other: Observational study exploring the epidemiology and outcomes of AKI in critical COVID-19 patients admitted to the ICU — Critical COVID-19 patients admitted to the ICU

SUMMARY:
The aim of this study is to evaluate the rate and outcomes of COVID-19 associated acute kidney injury (AKI) and use of kidney replacement therapy (KRT) in critically ill COVID-19 patients in ICUs in several large hospitals in Flanders, the northern region of Belgium. We will also explore the associations between several baseline risk factors for AKI, therapeutic strategies and COVID-19 related clinical signs and the occurrence of AKI and use of KRT.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the rate and outcomes of COVID-19 associated acute kidney injury (AKI) and use of kidney replacement therapy (KRT) in critically ill COVID-19 patients in ICUs in several large hospitals in Flanders, the northern region of Belgium. We will also explore the associations between several baseline risk factors for AKI, therapeutic strategies and COVID-19 related clinical signs and the occurrence of AKI and use of KRT.

This will be a cohort analysis of the rate of COVID-19 associated AKI and KRT during the period 1 February 2020 - 31 January 2021 in 6 large hospitals in Flanders Belgium and 3 Flemish University Hospitals. We will collect patients' baseline characteristics, specific treatment for COVID-19, other relevant therapies and severity of illness and ICU and hospital outcome data. AKI will be assessed during ICU stay up to 21 days of ICU stay, and will be defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) definition. In addition, we will assess occurrence of AKI stages, duration of AKI, duration of AKI integrated with severity stage of AKI into the area under the curve of AKI, occurrence of rapid reversal of AKI, occurrence of Acute Kidney Disease (AKD) defined according to KDIGO.

ELIGIBILITY:
Inclusion Criteria:

* Severe Acute Respiratory Syndrome CoronaVirus-2 (SARS-CoV-2) infection confirmed by Polymerase Chain Reaction (PCR) on nasopharyngeal swab or oropharyngeal swab or rectal swab or bronchoalveolar aspirate
* admission to the ICU for monitoring or organ support

Exclusion Criteria:

* asymptomatic COVID-19 patients admitted to the ICU for medical reason not related to COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive Critical COVID-19 patients admitted to the ICU
Sampling Method: Probability Sample
Enrollment: 1286 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | up to day 21 of ICU admission
  AKI occurrence and severity stages defined according to KDIGO
Kidney outcome | day 30 after ICU admission
  use of KRT and eGFR in patients without AKI (no AKI), AKI, and AKI stages
Mortality | day 30 after ICU admission
  Mortality of AKI and no AKI patients will be compared
Survival | AKI and AKD will be classified up to day 21 of ICU stay, and survival will be assessed up to day 30 or hospital discharge whichever is last
  Survival of no AKI, AKI and AKI stages, AKD, and rapid reversal up to day 30 or hospital discharge whichever comes last

SECONDARY OUTCOMES:
Acute Kidney Injury (AKI) creatinine criteria | up to day 21 of ICU admission
  AKI occurrence and severity stages defined according to KDIGO creatinine criteria
Acute Kidney Injury (AKI) urine output criteria | up to day 21 of ICU admission
  AKI occurrence and severity stages defined according to KDIGO urine output criteria
Acute Kidney Injury (AKI), rapid reversal | up to day 21 of ICU admission
  Occurrence of AKI for 48-h or less
Acute Kidney Disease (AKD) | up to day 21 of ICU admission
  Occurrence and severity staging of AKD according to KDIGO criteria
AKI-Area Under the Curve (AUC) | up to day 21 of ICU admission
  Assessment of AKI-AUC which is defined as the sum of the daily maximum severity stage of AKI
Mortality AKD | day 30 after ICU admission
  Mortality of patients with AKD and severity stages of AKD will be compared to no AKI and patients with AKI and different AKI stages
Mortality AKI rapid reversal | day 30 after ICU admission
  Mortality of patients with AKI rapid reversal ill be compared to no AKI and patients with AKI and different AKI stages
Mortality AKI stage 2-3 | day 30 after ICU admission
  Mortality of patients with AKI stage 2 or greater and patients with no AKI or AKI stage 1 will be compared
Mortality AKI treated with KRT | day 30 after ICU admission
  Mortality of patients with AKI treated with KRT and patients with no AKI or AKI stage 1, 2 or 3 will be compared
Mortality AKI creatinine criteria versus urine output criteria versus full KDIGO | day 30 after ICU admission
  Mortality of patients with AKI and patients with no AKI will be compared
Mortality AKI-AUC | day 30 after ICU admission
  Mortality of quartiles of AKI-AUC will be assessed
Kidney outcome AKI KDIGO creatinine or urine output | day 30 after ICU admission
  use of KRT and eGFR in no AKI, AKI on creatinine or urine output criteria and AKI stages, Rapid Reversal of AKI, and AKD and stages
Duration of AKI and AKD | up to day 21 of ICU admission
  Duration of AKI, AKI on creatinine or urine output criteria and AKI stages, Rapid Reversal of AKI, and AKD and stages
Survival AKI-AUC | AKI-AUC will be assessed up to day 21 of ICU stay, and survival will be assessed up to day 30 or hospital discharge whichever is last
  Survival up to day 30 or hospital discharge (whichever is last) for quartiles of AKI-AUC will be assessed
Recovery of AKI and AKD | day 30 after ICU admission
  Recovery of AKI, AKI stages, AKD and AKD stages, KRT will be assessed
Timing of AKI, AKI severity grades and use of KRT | ICU admission up to day 21
  timing of occurrence of AKI in relation to onset of symptoms, hospital admission, ICU admission
KRT modality | ICU admission up to day 21
  initial modality of KRT and anticoagulation used
use of KRT | ICU admission up to day 21
  number of KRT treatment days, and KRT free days
Subgroup analysis: Mechanical Ventilation | ICU admission up to day 21
  outcomes will be assessed in patients with and without mechanical ventilation at time of start of AKI
Subgroup analysis: Chronic Kidney Disease (CKD) (estimated glomerular filtration rate (eGFR)<60 mL/min) | ICU admission up to day 21
  outcomes will be assessed in patients with and without CKD as baseline kidney function
Subgroup analysis: elderly (>= 65 y) | ICU admission up to day 21
  outcomes will be assessed in patients older and younger than 65y
Subgroup analysis: obese (BMI>30 kg/m2) | ICU admission up to day 21
  outcomes will be assessed in obese patients and non-obese
Subgroup analysis: prone ventilation | ICU admission up to day 21
  outcomes will be assessed in patients treated with mechanical ventilation and in prone position
Subgroup analysis: extracorporeal membrane oxygenation (ECMO) | ICU admission up to day 21
  outcomes will be assessed in patients treated with ECMO

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, Md, PhD, Study Chair — University Hospital, Ghent; Greet De Vlieger, Md, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (9):
- Belgium (9):
  - UZ Antwerp, Antwerp
  - AZ St-Jan AV, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may propose additional analyses on the dataset. These proposals will be evaluated by the 2 study chairs Eric Hoste and Greet De Vlieger and the study group for eligibility

REFERENCES:
- [Background] Nadim MK, Forni LG, Mehta RL, Connor MJ Jr, Liu KD, Ostermann M, Rimmele T, Zarbock A, Bell S, Bihorac A, Cantaluppi V, Hoste E, Husain-Syed F, Germain MJ, Goldstein SL, Gupta S, Joannidis M, Kashani K, Koyner JL, Legrand M, Lumlertgul N, Mohan S, Pannu N, Peng Z, Perez-Fernandez XL, Pickkers P, Prowle J, Reis T, Srisawat N, Tolwani A, Vijayan A, Villa G, Yang L, Ronco C, Kellum JA. COVID-19-associated acute kidney injury: consensus report of the 25th Acute Disease Quality Initiative (ADQI) Workgroup. Nat Rev Nephrol. 2020 Dec;16(12):747-764. doi: 10.1038/s41581-020-00356-5. Epub 2020 Oct 15. PMID 33060844
- [Background] Ostermann M, Lumlertgul N, Forni LG, Hoste E. What every Intensivist should know about COVID-19 associated acute kidney injury. J Crit Care. 2020 Dec;60:91-95. doi: 10.1016/j.jcrc.2020.07.023. Epub 2020 Jul 28. PMID 32777758
- [Background] Chawla LS, Bellomo R, Bihorac A, Goldstein SL, Siew ED, Bagshaw SM, Bittleman D, Cruz D, Endre Z, Fitzgerald RL, Forni L, Kane-Gill SL, Hoste E, Koyner J, Liu KD, Macedo E, Mehta R, Murray P, Nadim M, Ostermann M, Palevsky PM, Pannu N, Rosner M, Wald R, Zarbock A, Ronco C, Kellum JA; Acute Disease Quality Initiative Workgroup 16.. Acute kidney disease and renal recovery: consensus report of the Acute Disease Quality Initiative (ADQI) 16 Workgroup. Nat Rev Nephrol. 2017 Apr;13(4):241-257. doi: 10.1038/nrneph.2017.2. Epub 2017 Feb 27. PMID 28239173
- [Background] Lameire NH, Levin A, Kellum JA, Cheung M, Jadoul M, Winkelmayer WC, Stevens PE; Conference Participants. Harmonizing acute and chronic kidney disease definition and classification: report of a Kidney Disease: Improving Global Outcomes (KDIGO) Consensus Conference. Kidney Int. 2021 Sep;100(3):516-526. doi: 10.1016/j.kint.2021.06.028. Epub 2021 Jul 9. PMID 34252450
- [Background] Ostermann M, Bellomo R, Burdmann EA, Doi K, Endre ZH, Goldstein SL, Kane-Gill SL, Liu KD, Prowle JR, Shaw AD, Srisawat N, Cheung M, Jadoul M, Winkelmayer WC, Kellum JA; Conference Participants. Controversies in acute kidney injury: conclusions from a Kidney Disease: Improving Global Outcomes (KDIGO) Conference. Kidney Int. 2020 Aug;98(2):294-309. doi: 10.1016/j.kint.2020.04.020. Epub 2020 Apr 26. PMID 32709292
- [Background] Hoste EA, Clermont G, Kersten A, Venkataraman R, Angus DC, De Bacquer D, Kellum JA. RIFLE criteria for acute kidney injury are associated with hospital mortality in critically ill patients: a cohort analysis. Crit Care. 2006;10(3):R73. doi: 10.1186/cc4915. Epub 2006 May 12. PMID 16696865
- [Derived] Schaubroeck H, Vandenberghe W, Boer W, Boonen E, Dewulf B, Bourgeois C, Dubois J, Dumoulin A, Fivez T, Gunst J, Hermans G, Lormans P, Meersseman P, Mesotten D, Stessel B, Vanhoof M, De Vlieger G, Hoste E. Acute kidney injury in critical COVID-19: a multicenter cohort analysis in seven large hospitals in Belgium. Crit Care. 2022 Jul 25;26(1):225. doi: 10.1186/s13054-022-04086-x. PMID 35879765